CLINICAL TRIAL: NCT04802356
Title: An Open Label, Multicenter, Phase II Study of Belantamab Mafodotin in Combination With VRd for the Treatment of Newly Diagnosed Transplant Eligible Multiple Myeloma Patients
Brief Title: Belantamab Mafodotin in Newly Diagnosed Transplant Eligible Multiple Myeloma Patients
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: PETHEMA Foundation (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GEM-BELA-VRd; 2020-002050-24 (EudraCT Number)
Record Dates: First submitted 2021-03-12; First posted 2021-03-17 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2025-11

CONDITIONS: Multiple Myeloma
Keywords: NEWLY DIAGNOSED; TRANSPLANT ELEGIBLE; BELANTAMAB MAFODOTIN
MeSH Terms: conditions — Multiple Myeloma | interventions — belantamab mafodotin; Bortezomib; Lenalidomide; Dexamethasone

STUDY DESIGN:
Intervention Model Description: This is a multicenter, open label, non-randomized single arm clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Multiple Myeloma experimental arm (Experimental): Combination of belantamab mafodotin + the combination treatment VRd (bortezomib, lenalidomide, dexamethasone)
  Interventions: Drug: Belantamab mafodotin; Drug: Bortezomib; Drug: Lenalidomide; Drug: Dexamethasone; Procedure: Autologous stem cell transplant (ASCT)

INTERVENTIONS:
Drug: Belantamab mafodotin — Dose of 2.5 mg/kg/every 8 weeks on day 1, intravenously, Induction: three induction cycles with belantamab mafodotin in combination with VRd.
  Consolidation: one cycle after 90 days of transplantation with belantamab mafodotin in combination with VRd.
  Maintenance: belantamab mafodotin in combination with lenalidomide until disease progression, patients withdrawal, death or up to two years, whichever occurs first
  Other Names: Blenrep
Drug: Bortezomib — Dose of 1.3 mg/m2, on days: 1, 4, 8 and 11 of every 28-day cycle. Subcutaneous administration Induction: 6 cycles Consolidation: 2 cycles
Drug: Lenalidomide — Dose of 25 mg/day on days 1-21 of every 28-day cycle. Oral administration. Induction: 6 cycles Consolidation: 2 cycles Maintenance: 10 mg/day on days 1-21 continuously (may increase up to 15 mg/day) until disease progression, patients withdrawal, death, whichever occurs first
Drug: Dexamethasone — Dose of 20 mg on days: 1, 2, 4, 5, 8, 9, 11 and 12 of every 28-day cycle. Oral administration Induction: 6 cycles Consolidation: 2 cycles
Procedure: Autologous stem cell transplant (ASCT) — High-dose melphalan (200 mg/m2) and ASCT will be performed as per routine practice

SUMMARY:
This is a multicenter, open label clinical trial evaluating the safety of the combination of belantamab mafodotin + the combination treatment VRd (bortezomib, lenalidomide, dexamethasone) in newly diagnosed (ND) transplant eligible multiple myeloma (MM) patients.

Eligible patients will be included in the study and they will receive three induction cycles with belantamab mafodotin (8-week cycles) and six induction cycles with VRd (4-week cycles). Immediately after the fourth VRd cycle, and in the absence of progression or unacceptable toxicity, mobilization of hematopoietic stem cells with G-CSF and subsequent apheresis will take place. Then, patients will receive one additional induction cycle with belantamab mafodotin (8-week cycle) and two additional induction cycles with VRd (4-week cycles) followed by intensification with high-dose melphalan (200mg/m2) and the autologous stem cell transplant. Three months after transplantation, and as long as clinical and hematological conditions allow, patients will receive one cycle of consolidation with belantamab mafodotin (8-week cycle) and two additional cycles of consolidation with VRd (4-week cycles) at the same doses as during induction and, subsequently, patients will receive maintenance treatment with lenalidomide (continuously until disease progression, patient withdrawal, unacceptable toxicity, loss to follow up, end of study or death) and belantamab mafodotin (for 2 years).

DETAILED DESCRIPTION:
This is a multicenter, open label clinical trial evaluating the safety of the combination of belantamab mafodotin + the combination treatment VRd (bortezomib, lenalidomide, dexamethasone) in newly diagnosed (ND) transplant eligible multiple myeloma (MM) patients.

The study comprise the following phases:

Induction: Cycles 1-6

Cycles will be of 8 weeks of duration for belantamab mafodotin and 28 days of duration for VRd:

* Belantamab mafodotin will be administered at the dose of 2.5 mg/kg/every 8 weeks on day 1, intravenously.
* Bortezomib will be given subcutaneously, at 1.3 mg/m2, on days: 1, 4, 8 and 11 of every 28-day cycle.
* Lenalidomide will be given as an oral drug, in the dose of 25 mg/day on days 1-21.
* Dexamethasone will be given as an oral drug, in the dose of 20 mg on days: 1, 2, 4, 5, 8, 9, 11 and 12.

Peripheral stem cell harvest will be performed after the fourth cycle of treatment to prevent mobilization failure.

Intensification with high-dose melphalan (200 mg/m2) and autologous stem cell transplant (ASCT) will be performed as per routine practice. Mobilization of hematopoietic stem cells (HSCs) will be carried out using high-dose G-CSF after the fourth induction cycle with VRd. The dose of G-CSF used will be at the discretion of each site according to the local rules. Apheresis will be initiated on day 4-5 of stimulation, once the number of CD34+ cells in peripheral blood have reached the minimum to proceed with the collection. The minimum number of CD34+ cells needed to carry out the transplant will be determined at the discretion of each site, although a minimum of 2 x106 CD34+/Kg is recommended, as well as cryopreservation, storage, defrosting and infusion of HSCs. If mobilization fails using G-CSF alone, the recommended action is to utilize plerixafor during the same procedure in order to save this time. Sites should administer plerixafor in accordance with their own established procedures. If this second attempt fails, the site can proceed to a third mobilization attempt using cyclophosphamide plus G-CSF.

Consolidation: Cycles 6-8

At day +90, after autologous stem cell transplant patients will receive consolidation treatment with 1 additional cycle of belantamab mafodotin + 2 additional cycles of VRd following the same scheme as in the induction:

* Belantamab mafodotin will be administered at the dose of 2.5 mg/kg/every 8 weeks on day 1, intravenously.
* Bortezomib will be given subcutaneously, at 1.3 mg/m2, on days: 1, 4, 8 and 11 of every 28-day cycle.
* Lenalidomide will be given as an oral drug, in the dose of 25 mg/day on days 1-21.
* Dexamethasone will be given as an oral drug, at the dose of 20 mg on days: 1, 2, 4, 5, 8, 9, 11 and 12 of every 28-day cycle.

Maintenance:

After completion of the consolidation treatment, all the responding patients will receive maintenance treatment with Lenalidomide (10 mg/day) + belantamab mafodotin (2.5 mg/kg/every 8 weeks, intravenously). Lenalidomide will be administered continuously until disease progression, patient withdrawal, unacceptable toxicity loss to follow up, end of study or death. Belantamab mafodotin will be administered for 2 years until disease progression, patient withdrawal, loss to follow up, unacceptable toxicity, end of study or death.

The trial has the following objectives:

Objectives:

Primary objective

● To evaluate the safety and tolerability of the combination of belantamab mafodotin + VRd in newly diagnosed transplant eligible multiple myeloma patients.

Secondary objectives ● To assess the efficacy of belantamab mafodotin in combination with VRd in terms of response rate focusing on complete response and MRD.

• Efficiency of hematopoietic stem cell collection after 2 induction cycles of treatment of belantamab mafodotin + 4 induction cycles of treatment of VRd.

ELIGIBILITY:
Inclusion Criteria:

1. Participant must have Newly diagnosed multiple myeloma. Newly diagnosed subjects must have symptomatic disease following the IMWG updated criteria (Rajkumar Lancet 2014, Appendix 6).
2. Participant must have a measurable secretory disease defined as either serum monoclonal protein of ≥ 0,5 g/dl or urine monoclonal (light chain) protein ≥ 200mg/24h.For patients whose disease is only measurable by serum FLC, the involved FLC should be ≥ 10mg/L (100 mg/dl), with an abnormal serum FLC ratio.
3. Newly diagnosed participants must be eligible for stem cell transplant at investigator criteria.
4. Participant must have an Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 2
5. Participant must be ≥ 18 years of age
6. Participant must have adequate organ function, defined as follows:

   System Laboratory Values Hematologic Absolute neutrophil count (ANC) ≥1.5 X 109/L Hemoglobin ≥8.0 g/dL Platelets ≥75 x 109/L for subjects in whom <50% of bone marrow nucleated cells are plasma cells; otherwise platelet count >50 × 109/L Calcium corrected serum calcium <14 mg/dL (<3.5 mmol/L); or free ionized calcium <6.5 mg/dL (<1.6 mmol/L); Hepatic Total bilirubin ≤1.5X ULN (Isolated bilirubin ≥1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%) ALT ≤2.5 X ULN AST ≤2.5 X ULN Renal eGFRa ≥30 mL/min/ 1.73 m2 Spot urine (albumin/creatinine ratios (spot urine) <500 mg/g (56 mg/mmol)
7. Female participants: contraceptive use should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.

   A female participant is eligible to participate if she is not pregnant or breastfeeding, and at least one of the following conditions applies:
   * Is not a woman of childbearing potential (WOCBP) OR
   * Is a WOCBP and using a contraceptive method that is highly effective (with a failure rate of <1% per year), preferably with low user dependency, during the intervention period and for at least 4 months after the last dose of study intervention and agrees not to donate eggs (ova, oocytes) for the purpose of reproduction during this period. The investigator should evaluate the effectiveness of the contraceptive method in relationship to the first dose of study intervention.

   A WOCBP must have a negative highly sensitive serum pregnancy test (as required by local regulations) within 72 hours before the first dose of study intervention and agree to use a highly effective method of contraception during the study and for 4 months after the last dose of belantamab mafodotin. Additional requirements for pregnancy testing during and after study intervention The investigator is responsible for review of medical history, menstrual history, and recent sexual activity to decrease the risk for inclusion of a woman with a nearly undetected pregnancy.

   Nonchildbearing potential is defined as follows (by other than medical reasons):
   * ≥45 years of age and has not had menses for >1 year
   * Patients who have been amenorrhoeic for <2 years without history of a hysterectomy and oophorectomy must have a follicle stimulating hormone value in the postmenopausal range upon screening evaluation Post-hysterectomy, post-bilateral oophorectomy, or post-tubal ligation. Documented hysterectomy or oophorectomy must be confirmed with medical records of the actual procedure or confirmed by an ultrasound. Tubal ligation must be confirmed with medical records of the actual procedure.
8. Male participants: contraceptive use should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.

   Male participants are eligible to participate if they agree to the following during the intervention period and for at least 6 months:
   * Refrain from donating sperm

   PLUS either:
   * Be abstinent from heterosexual intercourse as their preferred and usual lifestyle (abstinent on a long term and persistent basis) and agree to remain abstinent. OR
   * Must agree to use contraception/barrier as detailed below:

   Agree to use a male condom and female partner to use an additional highly effective contraceptive method with a failure rate of <1% per year as when having sexual intercourse with a woman of childbearing potential (including pregnant females). All prior treatment-related toxicities (defined by National Cancer Institute- Common Toxicity Criteria for Adverse Events (NCI-CTCAE), version 4.0 (must be ≤ Grade 1 at the time of enrolment except for alopecia).
9. Participant must be able to understand the study procedures and agree to participate in the study by providing written informed consent.

Exclusion Criteria:

Patients that present any of the following exclusion criteria cannot be included in the trial:

1. Participant has a diagnosis of primary amyloidosis, monoclonal gammopathy of undetermined significance (MGUS), smoldering multiple myeloma (SMM), plasma cell leukemia or active POEMS syndrome at the time of screening.
2. Participant has malignancies other than disease under study, except for any other malignancy from which the participant has been disease-free for more than 2 years and, in the opinion of the principal investigators, will not affect the evaluation of the effects of this clinical trial treatment on the currently targeted malignancy. Participants with curatively treated non-melanoma skin cancer may be enrolled.
3. Participant has meningeal involvement of multiple myeloma.
4. Pregnant or breastfeeding females.
5. Participant is simultaneously enrolled in other interventional clinical trial.
6. Participant must has used an investigational drug within 14 days or five half-lives, whichever is shorter, preceding the first dose of study drug.
7. Participant has used of any anti-myeloma drug therapy, except for steroid pulses in case of emergency (40 mg of dexamethasone for 4 days), the administration of bisphosphonates or antialgic radiotherapy or due to the presence of plasmacytomas requiring some emergency.
8. Participant who have received prior treatment with a monoclonal antibody within 30 days of receiving the first dose of study drugs.
9. Participant has a known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to: belantamab mafodotin, lenalidomide, boronic acid (bortezomib), dexamethasone or any of the components of the study treatment.
10. Participant who have had major surgery ≤ 4 weeks prior to initiating protocol therapy.
11. Participant who have current corneal epithelial disease except mild punctate keratopathy
12. Participant has peripheral neuropathy or neuropathic pain grade ≥2, as defined by the National Cancer Institute Terminology Criteria for Adverse Events (NCI CTCAE) Version 4.0 (APPENDIX 4).
13. Participant is unable or unwilling to undergone antithrombotic prophylactic treatment
14. Participant evidence of cardiovascular risk including any of the following:

    * Evidence of current clinically significant uncontrolled arrhythmias, including clinically significant ECG abnormalities such as 2nd degree (Type II) or 3rd degree atrioventricular (AV) block.
    * History of myocardial infarction, acute coronary syndromes (including unstable angina), coronary angioplasty, or stenting or bypass grafting within three months of Screening.
    * Class III or IV heart failure as defined by the New York Heart Association functional classification system [NYHA, 1994]
    * Uncontrolled hypertension
15. Incidence of gastrointestinal disease that may significantly alter the absorption of Lenalidomide.
16. Participant must not have current unstable liver or biliary disease defined by the presence of ascites, encephalopathy, coagulopathy, hypoalbuminemia, esophageal or gastric varices, persistent jaundice, or cirrhosis. Note: Stable chronic liver disease (including Gilbert's syndrome or asymptomatic gallstones) or hepatobiliary involvement of malignancy is acceptable if otherwise meets entry criteria
17. Presence of active renal condition (infection, requirement for dialysis or any other condition that could affect patient's safety). Participants with isolated proteinuria resulting from MM are eligible, provided they fulfil inclusion criteria
18. Participant who use contact lenses while participating in this study, except if contact lenses are removed during participation in the study
19. Participant who have had plasmapheresis within 7 days prior to first dose of study treatment.
20. Evidence of active mucosal or internal bleeding.
21. Any serious medical condition or psychiatric illness that would interfere in understanding of the informed consent form.
22. Uncontrolled endocrine diseases (i.e. diabetes mellitus, hypothyroidism or hyperthyroidism) (i.e. requiring relevant changes in medication within the last month, or hospital admission within the last 3 months).
23. Patients with acute diffuse infiltrative pulmonary disease and/or pericardial disease.
24. Patients with severe chronic obstructive pulmonary disease (COPD) or asthma with forced expiratory volume in the first minute (FEV1) less than 50%.
25. The subject is seropositive for human immunodeficiency virus (HIV) or presence of active hepatitis B infection (documented by a positive test for hepatitis B surface antigen [HBsAg], or hepatitis C (documented by a positive test for the surface antigen of hepatitis C [HCsAg] or positive quantification of HCV RNA Note: Participants with positive Hepatitis C antibody due to prior resolved disease can be enrolled, only if a confirmatory negative Hepatitis C RNA test is obtained.

Note: Hepatitis RNA testing is optional and participants with negative Hepatitis C antibody test are not required to also undergo Hepatitis C RNA testing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-04-07 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of deaths | Throughout the study period. Approximately 48 months
  Number of patients that are exitus after start of the study treatment
Incidence of adverse events (AEs) | Throughout the study period. Approximately 48 months
  Number of patients experiencing AEs, either treatment or non-treatment related, classified according to severity and graded according to NCTCAE V4.0
Incidence of analytical alterations | Throughout the study period. Approximately 48 months
  Changes in laboratory analytes from the hematology and blood chemistry panel after start of the study experimental treatment
Incidence of ocular events | Throughout the study period. Approximately 48 months
  Number of patients experiencing ocular alterations after start of the study experimental treatment.

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | Throughout the study period. Approximately 48 months
  The percentage of participants with a confirmed partial response (PR) or better (PR, Very good partial response (VGPR), Complete response (CR), stringent complete response (sCR)). Assessed Q4W during induction, three months after ASCT, after consolidation, q4W during maintenance until PD, unacceptable toxicity, death, withdrawal of consent, loss to follow-up or end of the study.
Complete Response Rate (CRR) | Throughout the study period. Approximately 48 months
  The percentage of participants with a confirmed complete response (CR) or better (stringent complete response (CR, sCR)). Assessed Q4W during induction, three months after ASCT, after consolidation, q4W during maintenance until PD, unacceptable toxicity, death, withdrawal of consent, loss to follow-up or end of the study.
Minimal Residual Disease (MRD) negativity rate | Throughout the study period. Approximately 48 months
  The percentage of participants who are MRD negative by next-generation flow cytometry (NGF). MRD will be evaluated after each phase of treatment (induction, autologous stem cell transplant, consolidation and once a year during maintenance). If there is suspect of CR at any time different of those previously specified, the MRD should be evaluated at the suspicion of CR. Assessed Q4W during induction, three months after ASCT, after consolidation, q4W during maintenance until PD, unacceptable toxicity, death, withdrawal of consent, loss to follow-up or end of the study.
Time to Response (TTR) | Throughout the study period. Approximately 48 months
  The time from the date of inclusion and the first documented evidence of response (PR or better) among participants who achieve confirmed PR or better.
Duration of Response (DoR) | Throughout the study period. Approximately 48 months
  The time from first documented evidence of PR or better until progressive disease (PD) or death due to PD among participants who achieved PR or better.
Progression-Free Survival (PFS) | Throughout the study period. Approximately 48 months
  The time from the date of inclusion until the earliest date of documented disease progression or death due to any cause.
Progression-Free Survival 2 (PFS2) | Throughout the study period. Approximately 48 months
  The time from inclusion to disease progression after initiation of new anti-cancer therapy or death from any cause, whichever is earlier. If disease progression after new anti-cancer therapy cannot be measured, a PFS event is defined as the date of discontinuation of new anti-cancer therapy, or death from any cause, whichever is earlier.
Overall Survival (OS) | Throughout the study period. Approximately 48 months
  Defined as the time from the date of inclusion until the date of death due to any cause.
Efficiency of hematopoietic stem cell collection | After cycle 4 of induction, 4 months after inclusion.
  Number of CD34 cells collected after 2 induction cycles of treatment of belantamab mafodotin + 4 induction cycles of treatment of VRd.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Victoria Mateos Manteca, M.D.; Ph.D., Study Chair — Hospital Universitario de Salamanca (Salamanca); Jesus San Miguel Izquierdo, M.D.; Ph.D., Study Chair — Clínica Universidad de Navarra (Pamplona)
Locations (14):
- Spain (14):
  - Hospital Son Llatzer, Palma de Mallorca, Balearic Islands
  - Hospital Universitario Marqués de Valdecilla, Santander, Cantabria
  - Hospital Universitario de Salamanca, Salamanca, Castille and León
  - Hospital Clínic I Provincial de Barcelona, Barcelona, Catalonia
  - Complejo Universitario Hospitalario de Santiago, Santiago de Compostela, Galicia
  - Hospital Gregorio Marañon, Madrid, Madrid
  - Hospital Universitario 12 de Octubre, Madrid, Madrid
  - Hospital de Cabueñes, Gijón, Principality of Asturias
  - Hospital Universitario de Canarias, San Cristóbal de La Laguna, Santa Cruz De Tenerife
  - Hospital Universitario y Policlínico de la Fe, Valencia, Valencia
  - Hospital Universitario de Gran Canaria Dr. Negrín, Las Palmas de Gran Canaria
  - Hospital Infanta Leonor, Madrid
  - Hospital General Universitario Morales Meseguer, Murcia
  - Hospital Virgen de la Arrixaca, Murcia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Darce JR, Arendt BK, Wu X, Jelinek DF. Regulated expression of BAFF-binding receptors during human B cell differentiation. J Immunol. 2007 Dec 1;179(11):7276-86. doi: 10.4049/jimmunol.179.11.7276. PMID 18025170
- [Background] Trudel S, Lendvai N, Popat R, Voorhees PM, Reeves B, Libby EN, Richardson PG, Hoos A, Gupta I, Bragulat V, He Z, Opalinska JB, Cohen AD. Antibody-drug conjugate, GSK2857916, in relapsed/refractory multiple myeloma: an update on safety and efficacy from dose expansion phase I study. Blood Cancer J. 2019 Mar 20;9(4):37. doi: 10.1038/s41408-019-0196-6. PMID 30894515
- [Background] Trudel S, Lendvai N, Popat R, Voorhees PM, Reeves B, Libby EN, Richardson PG, Anderson LD Jr, Sutherland HJ, Yong K, Hoos A, Gorczyca MM, Lahiri S, He Z, Austin DJ, Opalinska JB, Cohen AD. Targeting B-cell maturation antigen with GSK2857916 antibody-drug conjugate in relapsed or refractory multiple myeloma (BMA117159): a dose escalation and expansion phase 1 trial. Lancet Oncol. 2018 Dec;19(12):1641-1653. doi: 10.1016/S1470-2045(18)30576-X. Epub 2018 Nov 12. PMID 30442502
- [Background] Lonial S, Lee HC, Badros A, Trudel S, Nooka AK, Chari A, Abdallah AO, Callander N, Lendvai N, Sborov D, Suvannasankha A, Weisel K, Karlin L, Libby E, Arnulf B, Facon T, Hulin C, Kortum KM, Rodriguez-Otero P, Usmani SZ, Hari P, Baz R, Quach H, Moreau P, Voorhees PM, Gupta I, Hoos A, Zhi E, Baron J, Piontek T, Lewis E, Jewell RC, Dettman EJ, Popat R, Esposti SD, Opalinska J, Richardson P, Cohen AD. Belantamab mafodotin for relapsed or refractory multiple myeloma (DREAMM-2): a two-arm, randomised, open-label, phase 2 study. Lancet Oncol. 2020 Feb;21(2):207-221. doi: 10.1016/S1470-2045(19)30788-0. Epub 2019 Dec 16. PMID 31859245
- [Background] Cowan AJ, Allen C, Barac A, Basaleem H, Bensenor I, Curado MP, Foreman K, Gupta R, Harvey J, Hosgood HD, Jakovljevic M, Khader Y, Linn S, Lad D, Mantovani L, Nong VM, Mokdad A, Naghavi M, Postma M, Roshandel G, Shackelford K, Sisay M, Nguyen CT, Tran TT, Xuan BT, Ukwaja KN, Vollset SE, Weiderpass E, Libby EN, Fitzmaurice C. Global Burden of Multiple Myeloma: A Systematic Analysis for the Global Burden of Disease Study 2016. JAMA Oncol. 2018 Sep 1;4(9):1221-1227. doi: 10.1001/jamaoncol.2018.2128. PMID 29800065
- [Background] McCarthy PL, Holstein SA, Petrucci MT, Richardson PG, Hulin C, Tosi P, Bringhen S, Musto P, Anderson KC, Caillot D, Gay F, Moreau P, Marit G, Jung SH, Yu Z, Winograd B, Knight RD, Palumbo A, Attal M. Lenalidomide Maintenance After Autologous Stem-Cell Transplantation in Newly Diagnosed Multiple Myeloma: A Meta-Analysis. J Clin Oncol. 2017 Oct 10;35(29):3279-3289. doi: 10.1200/JCO.2017.72.6679. Epub 2017 Jul 25. PMID 28742454
- [Background] Attal M, Lauwers-Cances V, Hulin C, Leleu X, Caillot D, Escoffre M, Arnulf B, Macro M, Belhadj K, Garderet L, Roussel M, Payen C, Mathiot C, Fermand JP, Meuleman N, Rollet S, Maglio ME, Zeytoonjian AA, Weller EA, Munshi N, Anderson KC, Richardson PG, Facon T, Avet-Loiseau H, Harousseau JL, Moreau P; IFM 2009 Study. Lenalidomide, Bortezomib, and Dexamethasone with Transplantation for Myeloma. N Engl J Med. 2017 Apr 6;376(14):1311-1320. doi: 10.1056/NEJMoa1611750. PMID 28379796
- [Background] Durie BGM, Hoering A, Abidi MH, Rajkumar SV, Epstein J, Kahanic SP, Thakuri M, Reu F, Reynolds CM, Sexton R, Orlowski RZ, Barlogie B, Dispenzieri A. Bortezomib with lenalidomide and dexamethasone versus lenalidomide and dexamethasone alone in patients with newly diagnosed myeloma without intent for immediate autologous stem-cell transplant (SWOG S0777): a randomised, open-label, phase 3 trial. Lancet. 2017 Feb 4;389(10068):519-527. doi: 10.1016/S0140-6736(16)31594-X. Epub 2016 Dec 23. PMID 28017406
- [Background] Rosinol L, Oriol A, Rios R, Sureda A, Blanchard MJ, Hernandez MT, Martinez-Martinez R, Moraleda JM, Jarque I, Bargay J, Gironella M, de Arriba F, Palomera L, Gonzalez-Montes Y, Marti JM, Krsnik I, Arguinano JM, Gonzalez ME, Gonzalez AP, Casado LF, Lopez-Anglada L, Paiva B, Mateos MV, San Miguel JF, Lahuerta JJ, Blade J. Bortezomib, lenalidomide, and dexamethasone as induction therapy prior to autologous transplant in multiple myeloma. Blood. 2019 Oct 17;134(16):1337-1345. doi: 10.1182/blood.2019000241. PMID 31484647
- [Background] Kumar S, Paiva B, Anderson KC, Durie B, Landgren O, Moreau P, Munshi N, Lonial S, Blade J, Mateos MV, Dimopoulos M, Kastritis E, Boccadoro M, Orlowski R, Goldschmidt H, Spencer A, Hou J, Chng WJ, Usmani SZ, Zamagni E, Shimizu K, Jagannath S, Johnsen HE, Terpos E, Reiman A, Kyle RA, Sonneveld P, Richardson PG, McCarthy P, Ludwig H, Chen W, Cavo M, Harousseau JL, Lentzsch S, Hillengass J, Palumbo A, Orfao A, Rajkumar SV, Miguel JS, Avet-Loiseau H. International Myeloma Working Group consensus criteria for response and minimal residual disease assessment in multiple myeloma. Lancet Oncol. 2016 Aug;17(8):e328-e346. doi: 10.1016/S1470-2045(16)30206-6. PMID 27511158